CLINICAL TRIAL: NCT06563323
Title: A Single-arm Open-label Study Assessing Short-term (Week 6, 16) and Long-term (Week 32) Efficacy of Guselkumab in Adult Participants With Pyoderma Gangrenosum
Brief Title: Guselkumab in the Treatment of Adults With Pyoderma Gangrenosum (PG)
Acronym: GEORGE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); Ohio State University (Other)
Responsible Party: Principal Investigator, Alex Ortega Loayza, Doctor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Guselkumab for treatment of PG
Record Dates: First submitted 2024-08-07; First posted 2024-08-20 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Pyoderma Gangrenosum; Skin Diseases; Wound Heal; Pyoderma; Skin Ulcer
Keywords: Guselkumab; IL-23 Inhibitor
MeSH Terms: conditions — Pyoderma Gangrenosum; Skin Diseases; Pyoderma; Skin Ulcer | interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Guselkumab for PG (Experimental): Subjects with PG will be treated with 100 mg every 4 weeks of guselkumab for 28 weeks in addition to starting stable dose (at least 2 weeks) of prednisone at 20 mg daily. Prednisone will be tapered based on a pre-established algorithm assessed by investigator.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Subjects with PG will be treated with 100 mg in a pre-filled syringe to be injected subcutaneously every 4 weeks for 28 weeks.
  Other Names: Tremfya

SUMMARY:
A single-arm open-label study assessing short-term (week 6, 16) and long-term (week 32) efficacy of guselkumab in adult participants with pyoderma gangrenosum (PG)

DETAILED DESCRIPTION:
This is a Phase II study that will be open label and include a total of 17 patients who will receive the investigational product. PG will be defined by the investigator on the basis of results from clinical, histological and laboratory assessments. These patients will undergo 28 weeks of guselkumab dosed every 4 weeks and a stable dose of prednisone dosed daily with follow-up until week 40.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with study procedures/requirements
* Capable of giving informed consent
* Diagnosis of at least one PG ulcer by clinical, histological and laboratory assessments with a minimum wound size of 4 cm2.
* Undergoing at least once a week standard of care wound care at home or at a wound care facility
* Are candidate for systemic therapy. Must be on a stable dose of prednisone of 20 mg/day for at least two weeks prior to first drug administration.
* Males ages 18-99 who agree to not father a child or donate sperm while on study and at least 12 weeks following last dose of the study drug. If subject is sexually active male and could cause pregnancy, subject much be sure that female partner(s) are using birth control that works well or not have sex.
* Females ages 18-99; either of non-childbearing potential or of childbearing potential who test negative for pregnancy and agree to use at least two reliable methods of birth control or remain abstinent during the study for at least 12 weeks following the last dose of guselkumab.
* Willingness to travel to study site for all study visits or living >30 miles from study site and willing/able to participate in remote videoconferencing visits with access to a computer with internet and webcam capabilities.
* Be willing to undergo perilesional and non-lesional skin biopsy at week 0 and week 32 resulting in 4 biopsies during the course of the study. Participants can choose if they are willing to provide 2 additional biopsies at week 16. Refusal to give consent for any of the optional research samples does not exclude participant from participation in the study.

Exclusion Criteria:

* Has previously received at any time any therapeutic agent directly targeted to IL-23 including, but not limited to, guselkumab, risankizumab, tildrakuzumab, or mirikizumab
* Any drug treatment specifically for PG including but not limited to biologics (or biosimilar of), experimental antibodies, small molecules and oral immunosuppressives used within washout periods specified below, prior to first dose of study drug:

  1. 12 weeks for ustekinumab, ixekizumab, secukinumab, brodalumab;
  2. 8 weeks for infliximab;
  3. 6 weeks for adalimumab;
  4. 4 weeks for cyclosporine A, etanercept, inhibitors of the JAK/TYK pathway and PD4 inhibitors;
  5. 2 weeks for Calcineurin inhibitor topicals (including but not limited to pimecrolimus and tacrolimus) and other advanced topicals (including but not limited to roflumilast and tapinarof).

If not specified specifically, a time of 4 weeks or 5 half-lives of the drug (whichever is longer) prior to first drug administration.

* Intralesional corticosteroids within 4 weeks of screening.
* Active clinically infected ulcers. Individuals will be eligible for enrollment following completed treatment and resolution of infection. Antibiotics for wound superinfection are allowed.
* Immunomodulating medications for managing underlying comorbidities associated with PG, but not PG itself (e.g., for irritable bowel disease (IBD) or rheumatoid arthritis), are allowed as combination therapy except for Methotrexate (MTX) and Leflunomide which are allowed individually but not in combination.
* Concurrent skin disease that is deemed to interfere with assessment of ulcer.
* Have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly or a history of lymphoproliferative disease within 5 years before screening; or currently has a known malignancy or has a history of malignancy within 5 years before screening, with the exception of a nonmelanoma skin cancer that has been adequately treated with no evidence of recurrence for at least 3 months before the first study drug administration or cervical carcinoma in situ that has been treated with no evidence of recurrence for at least 3 months before the first study drug administration.
* Recent (within past 6 months) cerebrovascular accident, myocardial infarction, coronary stenting. Uncontrolled hypertension - confirmed systolic blood pressure >160 mmHg or diastolic blood pressure >100 mm Hg.
* Clinically significant (per investigator's judgement) drug or alcohol abuse within the last 6 months preceding the Baseline Visit.
* Has not fully recovered from major surgery (e.g., requiring general anesthesia and hospitalization) within 8 weeks before screening, or has such surgery planned during the time the participant is expected to participate in the study (40 weeks) which in the opinion of the investigator would pose an unacceptable risk to the subject.
* Presence of significant uncontrolled respiratory, hepatic, renal, endocrine, hematologic, neurologic, or neuropsychiatric disorders, or abnormal laboratory screening values that, in the opinion of the investigator, pose an unacceptable risk to the subject if participating in the study or of interfering with the interpretation of the data.
* Have clinical laboratory test results at screening that are outside the normal reference range of the population and are considered clinically significant, or have any of the following specific abnormalities: Neutrophil count <1500 cells/µL, Lymphocyte count <500 cells/µL, Platelet count <100,000 cells/µL, AST or ALT or alkaline phosphatase > 2 times the upper limit of normal, Hemoglobin <10 g/dL, Serum creatinine ≥1.5 mg/dL (SI: ≤137 μmol/L), White blood cells <3500 cells/ µL
* Participant has known allergies, hypersensitivity, or intolerance to guselkumab or its excipients.
* Individuals who are pregnant, lactating or breastfeeding.
* History of chronic or recurrent infections, or active, untreated, acute infection, or immunocompromised to an extent that participation in the study would pose an unacceptable risk to the subject based on the investigator's clinical assessment.
* Clinically serious infection or received intravenous antibiotics for an infection, within 8 weeks before first dose.
* Have signs or symptoms suggestive of active Tuberculosis (TB) upon medical history and/or physical examination. An exception is made for participants who are currently receiving treatment or will initiate treatment for latent TB prior to first administration of study intervention. For participants with a history of treated latent TB there must be documentation of appropriate treatment prior to the first administration of study intervention.
* Positive for human immunodeficiency virus (HIV), active hepatitis B virus, or hepatitis C virus. A positive Hepatitis B surface antibody test with a corresponding negative hepatitis B surface antigen test indicates immunity to the disease and will not be exclusionary.
* Symptomatic herpes zoster infection within 12 weeks of screening or recurrent or disseminated (even a single episode) herpes zoster.
* Symptomatic herpes simplex or disseminated (even a single episode) herpes simplex at the Week 0 (baseline) visit.
* History of disseminated opportunistic infections (e.g., listeriosis and histoplasmosis).
* Have received a live vaccine within 12 weeks prior to baseline or intend to have a live vaccine during the course of the study or 4 weeks after last study drug administration or 12 weeks after last study drug administration for Bacillus Calmette-Guérin (BCG) vaccine.
* Have any other condition that precludes the subject from following and completing the protocol, in the opinion of the investigator.
* Are investigator site personnel directly affiliated with this study and/or their immediate families (spouse, parent, child, or sibling).
* Are currently enrolled in, or discontinued from a clinical trial involving an investigational product or non-approved use of a drug or device within the last 4 weeks or a period of at least 5 half-lives of the last administration of the drug, whichever is longer, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-08-13 (Estimated); Study Completion 2027-08-13 (Estimated)

PRIMARY OUTCOMES:
Healing | Week 32
  Defined as the proportion of patients with complete re-epithelization, defined as a100% re-epithelialization without any drainage of the target ulcer at week 32.

SECONDARY OUTCOMES:
Physician Global Assessment (PGA) | Week 32
  Assessing the proportion of patients that show target ulcer healing in response to study treatment as measured by achieving PGA between 0 and 1 after treatment with guselkumab at week 32. This scale has been used in previous trials:
  0 = total resolution of target ulcer with no signs of active PG
  1= almost completely healed target ulcer with only minimal signs of active PG 2 = evidence of target ulcer healing which involves at least 50% of ulcer/ulcer margin 3 = evidence of target ulcer healing which involves less than 50% of ulcer/margin 4 = no evidence of target healing ulcer
Decrease in ulcer area size long-term | Week 32
  The proportion of patients with decrease in ulcer area size of at least 50% after treatment at week 32
Decrease in ulcer area size short-term | Week 16
  The proportion of patients with decrease in ulcer area size of at least 50% after treatment at Week 16
Mean decrease in ulcer area size short-term | Week 16
  Mean decrease in ulcer area size from Week 0 to Week 16
Mean decrease in ulcer area size long-term | Week 32
  Mean decrease in ulcer area size from Week 0 to Week 32
Skindex Mini | Week 32
  The Skindex Mini is a 3-item questionnaire, assessing symptom, emotion, and function related to skin disease. We will measure the mean change in Skindex Mini score from Week 0 to Week-32 will be reported with two-sided 95% confidence interval. Change in Skindex Mini score will be analyzed using a paired t-test with 0.05 significance level. Generalized estimating equation (GEE) methods will be further used to characterize changes in Skindex Mini score (max = 5, min = 0) over time. Higher scores indicated worsened quality of life due to skin disease.
Skin pain scale improvement over 7 days | Week 0 to 32
  The proportion of participants achieving a minimum of a 2 point decrease in the NRS at Week 0 and Week 32 The pain NRS is a subject-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable" in the last 7 days.
Skin pain scale improvement over 24 hours | Week 0 to 32
  The proportion of participants achieving an improvement in reported peak pain Numeric Rating Scale (NRS) assessment at Week 0 and Week 32. The peak pain NRS assessment is a subject-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable" in the last 24 hours
Change in physical function | Week 0 to 32
  The mean change in participant physical function from Week 0 to Week 32. Physical function is a subject-administered 5 category scale that assesses the impact of PG on participant physical function from "with no difficulty" to "can't do because of ulcer".
Mean change in global assessment score | Week 0 to 32
  The mean change in participant global assessment from Week 0 to Week 32. The participant global assessment is a subject administered 5 category scale (ranging from "clear" to "severe" that measures participant perspective of the status of their skin disease.
Target ulcer remains healed | Week 40
  The proportion of participants with target ulcer that remains healed by Week 40
Time to recurrence | Week 40
  Time to recurrence defined as the duration of time from documented target lesion healing and further episodes of PG at any site.
Treatment failure | Week 32
  The number of participants experiencing treatment failure.

OTHER OUTCOMES:
Evaluation of cytokine gene expression | Week 0 and Week 32
  Cytokine gene expression before and after treatment in skin, wound fluid, saliva and blood samples measured by enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Alex G Ortega-Loayza, MD, MCR, Principal Investigator — Oregon Health and Science University, Department of Dermatology
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ormerod AD, Thomas KS, Craig FE, Mitchell E, Greenlaw N, Norrie J, Mason JM, Walton S, Johnston GA, Williams HC; UK Dermatology Clinical Trials Network's STOP GAP Team. Comparison of the two most commonly used treatments for pyoderma gangrenosum: results of the STOP GAP randomised controlled trial. BMJ. 2015 Jun 12;350:h2958. doi: 10.1136/bmj.h2958. PMID 26071094
- [Background] Guillo L, D'Amico F, Danese S, Peyrin-Biroulet L. Ustekinumab for Extra-intestinal Manifestations of Inflammatory Bowel Disease: A Systematic Literature Review. J Crohns Colitis. 2021 Jul 5;15(7):1236-1243. doi: 10.1093/ecco-jcc/jjaa260. PMID 33367674
- [Background] Baier C, Barak O. Guselkumab as a treatment option for recalcitrant pyoderma gangrenosum. JAAD Case Rep. 2020 Dec 14;8:43-46. doi: 10.1016/j.jdcr.2020.12.005. eCollection 2021 Feb. No abstract available. PMID 33490346
- [Background] Burgdorf B, Schlott S, Ivanov IH, Dissemond J. Successful treatment of a refractory pyoderma gangrenosum with risankizumab. Int Wound J. 2020 Aug;17(4):1086-1088. doi: 10.1111/iwj.13359. Epub 2020 Apr 7. No abstract available. PMID 32266771
- [Background] Reese AM, Erickson K, Reed KB, Ortega-Loayza AG. Modified dose of guselkumab for treatment of pyoderma gangrenosum. JAAD Case Rep. 2022 Jan 6;21:38-42. doi: 10.1016/j.jdcr.2021.11.030. eCollection 2022 Mar. No abstract available. PMID 35146098
- [Background] Guenova E, Teske A, Fehrenbacher B, Hoerber S, Adamczyk A, Schaller M, Hoetzenecker W, Biedermann T. Interleukin 23 expression in pyoderma gangrenosum and targeted therapy with ustekinumab. Arch Dermatol. 2011 Oct;147(10):1203-5. doi: 10.1001/archdermatol.2011.168. Epub 2011 Jun 16. PMID 21680759
- [Background] Langrish CL, Chen Y, Blumenschein WM, Mattson J, Basham B, Sedgwick JD, McClanahan T, Kastelein RA, Cua DJ. IL-23 drives a pathogenic T cell population that induces autoimmune inflammation. J Exp Med. 2005 Jan 17;201(2):233-40. doi: 10.1084/jem.20041257. PMID 15657292
- [Background] Ortega-Loayza AG, Nugent WH, Lucero OM, Washington SL, Nunley JR, Walsh SW. Dysregulation of inflammatory gene expression in lesional and nonlesional skin of patients with pyoderma gangrenosum. Br J Dermatol. 2018 Jan;178(1):e35-e36. doi: 10.1111/bjd.15837. Epub 2017 Dec 5. No abstract available. PMID 28734003
- [Background] Abdo AIK, Tye GJ. Interleukin 23 and autoimmune diseases: current and possible future therapies. Inflamm Res. 2020 May;69(5):463-480. doi: 10.1007/s00011-020-01339-9. Epub 2020 Mar 25. PMID 32215665
- [Background] Cepeda MS, Africano JM, Polo R, Alcala R, Carr DB. What decline in pain intensity is meaningful to patients with acute pain? Pain. 2003 Sep;105(1-2):151-7. doi: 10.1016/s0304-3959(03)00176-3. PMID 14499431
- See also: A Study of Guselkumab in Participants With Moderately to Severely Active Crohn's Disease — https://ClinicalTrials.gov/show/NCT04397263
- See also: A Study of Guselkumab Subcutaneous Therapy in Participants With Moderately to Severely Active Crohn's Disease — https://ClinicalTrials.gov/show/NCT05197049
- See also: A Study of the Efficacy and Safety of Guselkumab in Participants With Moderately to Severely Active Crohn's Disease — https://clinicaltrials.gov/study/NCT03466411
- See also: Guselkumab in the Treatment of Pityriasis Rubra Pilaris — https://ClinicalTrials.gov/show/NCT03975153